CLINICAL TRIAL: NCT00873821
Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MK0941 After Multiple Daily Administration in Subjects With Type 2 Diabetes
Brief Title: A Pharmacokinetic Study of MK-0941 After Multiple Daily Doses in Subjects With Type 2 Diabetes (MK-0941-012)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0941-012; 2008_533
Record Dates: First submitted 2009-03-31; First posted 2009-04-02 (Estimated); Results first posted 2012-07-11 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 3-((6-(ethylsulfonyl)-3-pyridinyl)oxy)-5-(2-hydroxy-1-methylethoxy)-N-(1-methyl-1H-pyrazol-3-yl)benzamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): MK-0941
  Interventions: Drug: MK-0941
- 2 (Placebo Comparator): Placebo Comparator
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: MK-0941 — Part 1 (in house): MK-0941 twice daily on Days 1 through 13 before breakfast and dinner with 240 mL water. The starting dose on Day 1 was 10 mg tablets twice daily and titrated to a maximum dose of 60 mg twice daily through Day 9. The Day 9 dose was maintained throughout Day 13. Part 2 (at home): participants continued treatment for an additional 14 days with MK-0941 60 mg tablets (or maximum dose achieved in Part 1) twice daily, before meals with 240 mL of water.
  Arms: 1
Drug: Comparator: Placebo — Part 1 (in house): placebo twice daily on Days 1 through 13 before breakfast and dinner with 240 mL water. Part 2 (at home): participants continued treatment for an additional 14 days with placebo twice daily, before meals with 240 mL of water.
  Arms: 2

SUMMARY:
A study to test the pharmacokinetics after twice daily administration of MK-0941 or placebo in subjects with type 2 diabetes who have inadequate control on metformin.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a BMI < 42 kg/m2
* Subject is taking >1500 mg metformin per day for at least 8 weeks
* Subject has HbA1c value of 7.0% and < 11% at screening
* Subject is willing to follow AHA weight maintaining diet and exercise program
* Subject is a nonsmoker for at least 6 months

Exclusion Criteria:

* Subject has type 1 diabetes
* Subject has a history of stroke or chronic seizure
* Subject has a history of neoplastic disease
* Subject has a history of gastrointestinal, cardiovascular, blood, liver kidney, respiratory, immunological or genitourinary disorders or diseases
* Subject is currently taking 2 or more diabetes medications
* Subject has glaucoma or is blind
* If female, subject is pregnant or breastfeeding
* Subject consumes > 3 alcoholic beverages per day
* Subject has had major surgery or has donated blood in the last 4 weeks

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-12; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Part 1 (in house): placebo twice daily on Days 1 through 13 before breakfast and dinner with 240 mL water. Part 2 (at home): participants continued treatment for an additional 14 days with placebo twice daily, before meals with 240 mL of water.
Period: Overall Study
Arm/Group | MK-0941 | Placebo
Started | 22 | 22
Completed | 22 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-0941 | Placebo | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Customized [Number; unit: participants]
  37 to 70 years | 22 | 22 | 44
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 13 | 11 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Clinical Adverse Experience
Description: An adverse experience was defined as any unfavorable and unintended change in the structure or function of the body temporally associated with the use of study drug. Adverse experiences were collected using Medical Dictionary for Regulatory Activities (MedDRA) version 13.0.
Time Frame: 2 months
Population: All study participants
Measure: Number; unit: participants
Arm/Group | MK-0941 | Placebo
Number analyzed (Participants) | 22 | 22
participants | 18 | 16

2. Primary Outcome: Number of Participants With Any Laboratory Adverse Experience
Description: Laboratory adverse experiences were those related to changes in hematology, fasted blood chemistry, or urinalysis laboratory results. Adverse experiences were collected using MedDRA version 13.0.
Time Frame: 2 months
Population: All study participants
Measure: Number; unit: participants
Arm/Group | MK-0941 | Placebo
Number analyzed (Participants) | 22 | 22
participants | 3 | 1

3. Primary Outcome: Change From Baseline to Day 13 in Weighted Mean Plasma Glucose Concentration
Description: Weighted mean plasma glucose concentration was calculated as the 24-hour area under the plasma concentration-time curve divided by 24
Time Frame: Baseline (predose Day 1) to Day 13
Measure: Least Squares Mean (Standard Deviation); unit: mg/dL
Arm/Group | MK-0941 | Placebo
Number analyzed (Participants) | 22 | 22
mg/dL
  Baseline | 196.4 (47.6) [26.33 to 55.32] | 194.6 (35.3)
  Change from baseline to Day 13 | -56.4 (33.9) | -15.6 (30.0)
Statistical Analysis 1: Comparison: MK-0941 vs Placebo; Difference (placebo minus MK-0941) in change from baseline to Day 13; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 40.83, 95% CI 2-sided [26.33 to 55.32]

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | MK-0941 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 18/22 | 16/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MK-0941 (N=22) | Placebo (N=22)
Vision blurred (Eye disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 6 | 4
Dyspepsia (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 2 | 3
Vomiting (Gastrointestinal disorders) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Dizziness (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 6 | 6
Tremor (Nervous system disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication guidelines.